CLINICAL TRIAL: NCT01571115
Title: Effects of Resistance Physical Exercise in Patients With Chronic Primary
Brief Title: Effects of Resistance Physical Exercise in Patients With Chronic Primary Insomnia
Acronym: IER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Marco Tulio de Mello, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 0147/11
Record Dates: First submitted 2012-03-21; First posted 2012-04-04 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Insomnia
Keywords: insomnia; resistance physical exercise; stretching
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Insomnia Stretching Exercise (Active Comparator): This group will realize stretching exercise
  Interventions: Behavioral: Physical Exercise
- Control (No Intervention): This group will not realize any type of intervention.
- Insomnia Physical Exercise (Active Comparator): This group will realize resistance physical exercise
  Interventions: Behavioral: Physical Exercise

INTERVENTIONS:
Behavioral: Physical Exercise
  Arms: Insomnia Physical Exercise; Insomnia Stretching Exercise

SUMMARY:
INTRODUCTION: The primary insomnia, according to the concepts of the DSM IV, is a disorder characterized by difficulty initiating or maintaining sleep, waking early or by non-restorative sleep, resulting in losses in the daily functioning of patients, such as lack of attention, concentration and memory, fatigue, moodiness and irritability that are potentially associated with changes in sleep architecture, especially the reduction in slow-wave sleep. The most widely used therapy for the treatment of insomnia is the drug, but currently the resistive exercise is an important non-pharmacological intervention known to provide enough increase in slow wave sleep, and improve other parameters of sleep, as well as reducing symptoms of anxiety that are directly associated with the framework of insomnia. OBJECTIVE: To evaluate the effect of chronic resistive exercise in sleep patterns, the profile of mood and quality of life of patients with chronic primary insomnia. METHODOLOGY: 30 patients will be selected (male and female) with chronic primary insomnia. (Clinical diagnosis based on DSM-IV) referred for ambulatory sleep disorders Sleep Institute - AFIP. The protocol will be conducted at the Center for Psychobiology and Exercise (CEPE) of the AFIP and the Sleep Institute. Volunteers will be randomized into 2 groups of 15 participants, which will hold a resistive exercise and the other stretching exercise. This study will consist of three assessments: Pre-intervention (baseline), intermediate Rating (2 months) and post-intervention (at the end of 4 months). In the program of resistive exercise will be held 48 sessions that involve upper and lower limbs, abdominal and paraspinal region. It will be initially used a relative intensity 50% 1-RM. After 2 months of training intensity will be increased to 60% of 1-RM. Each exercise will be conducted in three sets of 12 repetitions, at intervals of 30 seconds between sets and one minute between each exercise. The total duration of the training session will be approximately 50 minutes. Before starting the training, participants will hold for 5 minutes stretching and warming on a bicycle ergometer (Life Cycle 9100) or treadmill (Life Fitness 9100) for the same period. After the session, the volunteers performed repeated stretches at the start of training. The group submitted to follow the practice of stretching protocol performed by Tworoger et al. that consist of 48 sessions of stretching for 60 minutes of low intensity, three times a week. The session will begin with 5 minutes of walking around the room, followed by 45 minutes of stretching exercises that involve the upper and lower limbs, 8 to 10 types for each region and end with 10 minutes of relaxation. STATISTICAL ANALYSIS: The variables of sleep, body composition and maximal repetition test will be analyzed using the software Statistica 7.0 (StaSoft, INC). The appropriate statistical test, parametric or nonparametric, will be chosen according to the data of the sample groups.

DETAILED DESCRIPTION:
METHODOLOGY: 30 patients will be selected (male and female) with chronic primary insomnia. (Clinical diagnosis based on DSM-IV) referred for ambulatory sleep disorders Sleep Institute - AFIP. The protocol will be conducted at the Center for Psychobiology and Exercise (CEPE) of the AFIP and the Sleep Institute. Each patient will undergo an initial interview that will aim to clarify the objectives and procedures of the protocol, as well as obtaining the signature of the Consent for Participation in Research. During the interview, a questionnaire will be applied (Sleep Quality Index in Pittsburgh) (68) for assessment of subjective sleep complaints and depression scale (Beck Depression Inventory, BDI) (69). Then the patient will be submitted to general clinical examination, blood collection and conduct examinations and resting electrocardiograms. Later, it will be subjected to a polysomnographic procedures. Volunteers will be randomized into 3 groups of 10 participants, which will hold a resistive exercise and the other stretching exercise and other will be a control group. Inclusion criteria are: age between 30 and 55 years, clinical diagnosis of primary insomnia (DSM-IV, ICSD, 2005), complaints of insomnia for a period longer than 6 months and have at least one day complaining of prejudice resulting from insomnia (such as moodiness, irritability and/or cognitive impairment). The non-inclusion criteria are: the use of psychoactive drugs, history of psychiatric disorders, shift workers, people with other sleep disorders and/or depression, significant abnormalities in laboratory tests and clinical trials have apnea/hypopnea index - AHI> 15, present rate of periodic leg movements - IMPP> 15, show abnormalities in heart tests (resting and exercise ECG) and blood that might impede the practice of physical exercises and practice regular physical exercise. This study will consist of three assessments: Pre-intervention (baseline), intermediate Rating (2 months) and post-intervention (at the end of 4 months). In each evaluation the volunteers must attend the lab of CEPE to achieve the following: blood collection, will be carried out in fast, always in the morning, body composition assessment, will be performed later to collect blood, a repeat maximum test - 1RM - only group that is performing the exercise resistance, actigraphy and sleep diary (15 days); polysomnographic studies and questionnaires. In the program of resistive exercise will be held 48 sessions that involve upper and lower limbs, abdominal and paraspinal region. There will be 4 exercises for upper limb: biceps, triceps, back and chest; 4 for the lower limbs: flexors, extensors, abductors and adductors, an exercise in trunk flexion to the region of the abdomen and an extension to the paravertebral trunk. It will be initially used a relative intensity 50% 1-RM. After 2 months of training intensity will be increased to 60% of 1-RM. Each exercise will be conducted in three sets of 12 repetitions, at intervals of 30 seconds between sets and one minute between each exercise. The total duration of the training session will be approximately 50 minutes. Before starting the training, participants will hold for 5 minutes stretching and warming on a bicycle ergometer (Life Cycle 9100) or treadmill (Life Fitness 9100) for the same period. After the session, the volunteers performed repeated stretches at the start of training. The group submitted to follow the practice of stretching protocol performed by Tworoger et al. that consist of 48 sessions of stretching for 60 minutes of low intensity, three times a week. The session will begin with 5 minutes of walking around the room, followed by 45 minutes of stretching exercises that involve the upper and lower limbs, 8 to 10 types for each region and end with 10 minutes of relaxation.

ELIGIBILITY:
Inclusion Criteria:

* age between 30 and 55 years,
* clinical diagnosis of primary insomnia (DSM-IV, ICSD, 2005),
* complaints of insomnia for a period longer than 6 months and have at least one day complaining of prejudice resulting from insomnia (such as moodiness, irritability and/or cognitive impairment)

Exclusion Criteria:

* the use of psychoactive drugs,
* history of psychiatric disorders, shift workers,
* people with other sleep disorders and/or depression,
* significant abnormalities in laboratory tests and clinical trials have apnea/hypopnea index
* AHI > 15,
* present rate of periodic leg movements
* IMPP > 15,
* show abnormalities in heart tests (resting and exercise ECG) and blood that might impede the practice of physical exercises and practice regular physical exercise.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Baseline | Pre-intervention
  In each evaluation the volunteers must attend the lab of CEPE to achieve the following: blood collection, will be carried out in fast, always in the morning, body composition assessment, will be performed later to collect blood, a repeat maximum test - 1RM - only group that is performing the exercise resistance, actigraphy and sleep diary (15 days); polysomnographic studies and questionnaires.

SECONDARY OUTCOMES:
Intermediate Rating | After 2 months
  n each evaluation the volunteers must attend the lab of CEPE to achieve the following: blood collection, will be carried out in fast, always in the morning, body composition assessment, will be performed later to collect blood, a repeat maximum test - 1RM - only group that is performing the exercise resistance; polysomnographic studies and questionnaires.
Post-Intervention | After 4 months
  In each evaluation the volunteers must attend the lab of CEPE to achieve the following: blood collection, will be carried out in fast, always in the morning, body composition assessment, will be performed later to collect blood, actigraphy and sleep diary (15 days); polysomnographic studies and questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Túlio de Mello, Principal Investigator — Universidade Federal do Estado de São Paulo
Locations (1):
- Centro de Estudos em Psicobiologia e Exercicio, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Passos GS, Poyares D, Santana MG, D'Aurea CV, Youngstedt SD, Tufik S, de Mello MT. Effects of moderate aerobic exercise training on chronic primary insomnia. Sleep Med. 2011 Dec;12(10):1018-27. doi: 10.1016/j.sleep.2011.02.007. Epub 2011 Oct 22. PMID 22019457
- [Result] Reid KJ, Baron KG, Lu B, Naylor E, Wolfe L, Zee PC. Aerobic exercise improves self-reported sleep and quality of life in older adults with insomnia. Sleep Med. 2010 Oct;11(9):934-40. doi: 10.1016/j.sleep.2010.04.014. Epub 2010 Sep 1. PMID 20813580
- [Result] Passos GS, Poyares D, Santana MG, Garbuio SA, Tufik S, Mello MT. Effect of acute physical exercise on patients with chronic primary insomnia. J Clin Sleep Med. 2010 Jun 15;6(3):270-5. PMID 20572421
- [Derived] D'Aurea CVR, Poyares D, Passos GS, Santana MG, Youngstedt SD, Souza AA, Bicudo J, Tufik S, de Mello MT. Effects of resistance exercise training and stretching on chronic insomnia. Braz J Psychiatry. 2019 Jan-Feb;41(1):51-57. doi: 10.1590/1516-4446-2018-0030. Epub 2018 Oct 11. PMID 30328967